CLINICAL TRIAL: NCT02059954
Title: Vaginal Hysterectomy Versus Total Laparoscopic Hysterectomy for Benign Indications: A Randomized Controlled Trial
Brief Title: Vaginal vs. Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Collaborators: Austrian Urogynecology Working Group (AUWG) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26-122 ex 13/14; MUG 26-122 ex 13/14 (Other: MUGraz)
Record Dates: First submitted 2014-02-10; First posted 2014-02-11 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Uterine Fibroids; Uterine Leiomyoma; Abnormal Uterine Bleeding, Unspecified
Keywords: Hysterectomy
MeSH Terms: conditions — Leiomyoma; Myofibroma; Metrorrhagia | interventions — Hysterectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vaginal hysterectomy (Active Comparator): Vaginal hysterectomy
  Interventions: Procedure: Hysterectomy
- Total laparoscopic hysterectomy (Active Comparator): Laparoscopic hysterectomy
  Interventions: Procedure: Hysterectomy

INTERVENTIONS:
Procedure: Hysterectomy

SUMMARY:
Hysterectomy for benign indication is one of the most common surgical procedures in women. Numerous reviews and guidelines recommend the vaginal approach for benign hysterectomy, but the proportion of laparoscopic (and robotic) hysterectomies is increasing.

This study will compare a range of clinical and subjective outcomes of vaginal vs. total laparoscopic hysterectomy. Outcomes include operating time, postoperative recovery, return to work as well as cosmesis, quality of life and sexual health.

ELIGIBILITY:
Inclusion Criteria:

* benign indication for vaginal hysterectomy (e.g., abnormal uterine bleeding, fibroids, atypical endometrial hyperplasia)
* clinical exam indicates vaginal hysterectomy is feasible
* no major concomitant surgery
* able to complete questionnaires in German

Exclusion Criteria:

* uterine malignancy
* major concomitant surgery (e.g., for incontinence or prolapse)
* clinical exam indicating vaginal hysterectomy not feasible
* contraindication for surgery or laparoscopy

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Operating time (min.) | Surgery
  Operating time (min.)

SECONDARY OUTCOMES:
Complications | 6 weeks
  Intraoperative and postoperative complications
Anesthesia time (min.) | surgery
Quality of life | 12 months
Sexual health | 12 months
Return to work | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karl F Tamussino, MD, Study Chair — Medical University of Graz; Rene W Laky, MD, Principal Investigator — Medical University of Graz
Locations (3):
- Austria (3):
  - Krankenhaus der Barmherzigen Brüder, Abteilung Gynäkologie, Graz
  - Medical University of Graz/Dept. OB/GYN, Graz
  - LKH Leoben/Abteilung Gynäkologie, Leoben